CLINICAL TRIAL: NCT02204696
Title: The Role of Tonsillectomy in Adults With Marked Tonsillar Hypertrophy and Obstructive Sleep Apnea
Brief Title: Tonsillectomy in Adults With Tonsillar Hypertrophy and Obstructive Sleep Apnea
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: University of Southern California (Other)
Collaborators: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Eric Kezirian, Professor, University of Southern California
Other Study IDs: HS-13-00794
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; obstructive sleep apnea; sleepiness; quality of life
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Sleepiness | interventions — Tonsillectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tonsillectomy: All participants will undergo baseline sleep study, a second preoperative sleep study after a period of watchful waiting, and a postoperative sleep study.
  Interventions: Procedure: Tonsillectomy

INTERVENTIONS:
Procedure: Tonsillectomy — Study participants will be scheduled for tonsillectomy based on clinical indications, with the need for surgery determined prior to study enrollment and not based on study enrollment.

SUMMARY:
The purpose of the study is to determine if tonsillectomy eliminates symptoms of obstructive sleep apnea in patients with obstructive sleep apnea and marked tonsillar hypertrophy with normal soft palate and uvula length.

DETAILED DESCRIPTION:
Purpose: To determine if tonsillectomy eliminates symptoms of obstructive sleep apnea in patients with obstructive sleep apnea and marked tonsillar hypertrophy with normal soft palate and uvula length.

Specific Aims: 1. To determine if tonsillectomy eliminates obstructive sleep apnea as determined by polysomnography. 2. To determine if tonsillectomy eliminates excessive daytime sleepiness and other obstructive sleep apnea symptoms.

Rationale: Current surgical procedures for obstructive sleep apnea include tonsillectomy with soft palate surgery (including uvulopalatopharyngoplasty). Tonsillectomy alone may provide sufficient benefit in adults with marked tonsillar hypertrophy and normal soft palate and uvula length, avoiding the need for additional soft palate surgery.

Intervention: Tonsillectomy will be performed as standard of care, in patients who would be undergoing said surgery regardless of study. Study intervention includes multiple home sleep studies to determine effect of tonsillectomy in impacting symptoms of sleep apnea.

Study Population: Inclusion criteria: Subjects must be at least 18 years old, have documented obstructive sleep apnea; be willing to undergo 3 home sleep studies; and have markedly hypertrophic (3+ or 4+) tonsils. Exclusion criteria: Subjects must not have any craniofacial abnormality; normal soft palate length (<4 cm) and uvula length ((<2 cm); must have no history of chronic obstructive pulmonary disease, untreated psychological disorder, restless leg syndrome, alcohol or drug abuse; must have a body mass index <35; must not plan to use continuous positive airway pressure during the study period, and lack significant nasal obstruction. The subjects will serve as their own control.

Methods and Follow Up: This two-center prospective study will include evaluation of demographics, clinical symptoms, extent of tonsillar hypertrophy, sleep habits, and home sleep studies. All subjects will undergo a 4-8 week period of watchful waiting (standard minimum delay for scheduling surgery), followed by tonsillectomy alone, with values at baseline compared to a period of watchful waiting and post-tonsillectomy.

Outcomes: Primary outcome is apnea-hypopnea index (from home sleep study). Exploratory outcomes include other sleep study results and subjective assessments (sleep-related quality of life with the Functional Outcome of Sleep Questionnaire and daytime sleepiness with the Epworth Sleepiness Scale).

Statistics and Plans for Analysis: The minimum sample size is 44 subjects, with an enrollment target of 60 subjects that will accommodate a 25% dropout rate. Standard statistical tests (e.g., paired t-tests for continuous measures) will evaluate potential differences between outcome measures at baseline vs. post-watchful waiting and baseline vs. post-tonsillectomy. Similarly, standard and appropriate statistical tests (e.g, t-tests for continuous measures) will compare changes with watchful waiting vs. tonsillectomy (e.g., baseline vs. post-watchful against baseline vs. post-tonsillectomy).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Documented obstructive sleep apnea (with central apneas of the total number of apneas plus hypopneas)
* Able to complete all forms in English and follow-up appointments
* Willing to undergo 3 home sleep studies; and markedly hypertrophic (3+ or 4+) tonsils
* Tonsil size of 3+ or 4+ corresponds to tonsils that occupy more than 50% of the space between the tonsillar fossa (side of the throat) and midline

Exclusion Criteria:

* No craniofacial abnormality
* No history of COPD, untreated psychological disorder, other sleep disorder, alcohol or drug abuse
* Body mass index <35 kg/m2
* Unable to tolerate other treatments for obstructive sleep apnea
* Soft palate length > 4 cm
* Uvula length > 2 cm
* No significant nasal obstruction

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with obstructive sleep apnea and tonsillar hypertrophy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
apnea-hypopnea index | 8 weeks
  This will be determined by home sleep study.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale score | 8 weeks
  This measure of daytime sleepiness will be assessed by questionnaire.
Functional Outcomes of Sleep Questionnaire score | 8 weeks
  This measure of sleep-related quality of life will be assessed by questionnaire.

OTHER OUTCOMES:
Insomnia Severity Index | 8 weeks
  This measure of insomnia severity will be assessed by questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Keck Hospital of USC, Los Angeles, California, United States